CLINICAL TRIAL: NCT04847635
Title: Subthreshold Laser Treatment for Reticular Pseudodrusen Secondary to Age-related Macular Degeneration
Acronym: PASCAL-RPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Fondazione G.B. Bietti, IRCCS (Other); University of Genova (Other); University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Querques Giuseppe, Head of Medical Retina & Imaging Unit, Clinical Professor, and Principal Investigator, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PASCAL-RPD
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Macular Degeneration, Senile; Laser Burn of Retina; Macular Degeneration Intermediate; Macular Degeneration, Dry
Keywords: Retina; Age-related macular degeneration; Reticular pseudodrusen; Sub-threshold laser
MeSH Terms: conditions — Macular Degeneration, Age-Related, 2; Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, longitudinal, interventional study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subthreshold laser group (Experimental): To evaluate the efficacy of Subthreshold laser in the treatment of reticular pseudodrusen.
  Interventions: Device: Pascal Synthesis 577 sub-threshold laser (Topcon Corporation, Tokyo, Japan)
- Sham group (Sham Comparator): The light from the retinal illumination system on the laser device will be used instead of the laser beam in all follow-up evaluations.
  Interventions: Device: Pascal Synthesis 577 sham (Topcon Corporation, Tokyo, Japan)

INTERVENTIONS:
Device: Pascal Synthesis 577 sub-threshold laser (Topcon Corporation, Tokyo, Japan) — The subthreshold laser treatment will be performed using subthreshold laser Pascal Synthesis 577 on a customized macular area.
  Arms: Subthreshold laser group
Device: Pascal Synthesis 577 sham (Topcon Corporation, Tokyo, Japan) — The laser treatment will be performed without any power (only the light beam) using subthreshold laser Pascal Synthesis 577 on a customized macular area.
  Arms: Sham group

SUMMARY:
Prospective, randomized, controlled, longitudinal, interventional multicentric study involving patients with reticular pseudodrusen secondary to AMD.

The objective of this study is to establish the effectiveness of subthreshold laser treatment in increase/prevent the decrease of the retinal sensibility in patients with reticular pseudodrusen, and to reduce the progression of RPD to atrophy.

Approximately 50 naïve patients with reticular pseudodrusen who underwent subthreshold laser treatment in perifoveal area. These patients should be randomized in the 2 study arms of the study. Patients will be evaluated at Screening/Baseline and then revaluated and retreated at month 3, 6 and 9. At month 12, all patients will be evaluated with a full ocular examination, visual acuity measurement (VA), optical coherence tomography (OCT) with autofluorescence, OCT-angiography and microperimetry.

The rationale of the study is to prevent the evolution of reticular pseudodrusen to atrophic degeneration.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* Presence of RPD secondary to AMD
* Best-corrected visual acuity (BCVA) between 20/20 and 20/400 inclusive
* Clear ocular media
* Ability to provide informed consent and attend all study visits

Exclusion Criteria:

* Presence of Geographic Atrophy (GA)
* Evidence of choroidal neovascularization in either eye
* Any prior treatment for AMD, aside from antioxidants
* Any corneal opacity, cataract formation and hemorrhage in the vitreous body, which may interfere with viewing by the laser surgeon of the target structures
* Aphakic eye with vitreous in the anterior chamber
* Neovascular Glaucoma
* Glaucoma caused by congenital angle anomalies
* Open angle of less than 90º or extensive peripheral anterior and low synechia, present circumferentially around the corner
* Significant corneal edema or reduced water clarity that obscures the view angle in detail
* Glaucoma secondary to active uveitis
* Any other ocular condition that would progress in the study period and confound visual acuity assessment
* Any ocular or systemic medication known to be toxic to the lens, retina or optic nerve Presence of idiopathic or autoimmune-associated uveitis
* Any intraocular surgery 3 months of entry
* Any prior thermal laser in the macula
* History of vitrectomy, filtering surgery, corneal transplant or retinal detachment surgery
* Previous therapeutic radiation in the ocular region in either eye
* Any treatment with an investigational agent in the previous 60 days before study entry
* Women of child-bearing potential, defined as all women less than 1 year postmenopausal or less than 6 weeks since sterilization (further definition can be found in Section 12.7) at Baseline, unless they are using highly effective methods of contraception during dosing of study treatment.
* Participation in an investigational drug, biologic, or device study within 6 Months prior to Baseline [Note: observational clinical studies solely involving over-the-counter vitamins, supplements, or diets are not exclusionary

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the retinal sensitivity - 12 months | 12 months
  Functional changes in the retinal sensitivity on customized microperimetry from day 0 to month 12 (unit of measure: dB)
Anatomical changes using structural optical coherence tomography (OCT) | 12 months
  Anatomical changes will be evaluated with retinal thickness (unit of measure: microns)
Rate of Progression | 12 months
  Rate of progression to advance AMD (GA and/or neovascular AMD)

SECONDARY OUTCOMES:
Changes in the retinal sensitivity - 6 months | 6 months
  Functional changes in the retinal sensitivity on customized microperimetry from day 0 to month 6 (unit of measure: dB)
Anatomical changes using fundus autofluorescence (FAF) | 12 months
  Anatomical changes will be evaluated analyzing the development of geographic atrophy using FAF
Genetic influence (% of AMD-associated single-nucleotide polymorphism (SNP) in treated patients) | 12 months
  The % of AMD-associated single-nucleotide polymorphism (SNP) will be evaluated analyzing the % of patients with an AMD-associated SNP in patients showing no progression vs progression to advance AMD (main outcome 3).
Anatomical changes using OCT-angiography (OCT-A) | 12 months
  Anatomical changes will be evaluated analyzing the perfusion density by means of OCT-A

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Massimo Nicolò, Genova
  - Giuseppe Querques, Milan
  - Mariacristina Parravano, Rome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Querques G, Sacconi R, Gelormini F, Borrelli E, Prascina F, Zucchiatti I, Querques L, Bandello F. Subthreshold laser treatment for reticular pseudodrusen secondary to age-related macular degeneration. Sci Rep. 2021 Jan 26;11(1):2193. doi: 10.1038/s41598-021-81810-7. PMID 33500505